CLINICAL TRIAL: NCT04418544
Title: Testing of Soniphi Vocal Feature Analysis Algorithm for COVID-19
Brief Title: Vocal Feature Analysis Algorithm for COVID-19 Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soniphi LLC (Industry)
Collaborators: UserWise, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 002 Soniphi
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Control: Do not test positive for COVID
  Interventions: Device: Device used to record voice for screening
- COVID-19 Positive: Test positive for Covid using swab test.
  Interventions: Device: Device used to record voice for screening

INTERVENTIONS:
Device: Device used to record voice for screening — voice recording

SUMMARY:
This is an observational, prospective, non-randomized, non-significant risk study collecting voice recordings from subjects who are being tested for COVID-19 by laboratory analysis of specimens obtained by nasal or naso-pharyngeal (NP) swab. Patients record their voices through an app on their mobile phone. Patients and health care providers will be blinded to the swab test results during Phase 2 of the study.

DETAILED DESCRIPTION:
The primary objective of this observational study is to determine if the Vocal Feature Analysis (VFA) Algorithm developed by Soniphi can screen for the COVID-19 condition from voice recordings. Patients eligible for the study are those being tested for COVID-19 based on molecular diagnostic testing of specimens obtained by nasal or nasopharyngeal swab.

No clinical decisions will be based on the recordings. The results of the algorithm analysis will not be made available to the subjects or their healthcare providers during or after the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged > 18 years
2. Provide a valid electronic informed consent form
3. Eligible patients are those meeting SOC guidelines for swab tests for COVID-19 and those providing an evaluable sample.
4. Stated willingness to provide evidence of their lab test results
5. Pregnant or lactating women may participate

Exclusion Criteria:

1. Presence of tracheostomy or past tracheostomy with permanent change to the voice due complications that involved the vocal cords.
2. Prior surgery which may influence the vocal cords, e.g., laryngeal, tracheal or esophageal surgery
3. Prior head, neck or throat cancer treated with radical neck dissection and/or radiation therapy that may influence the vocal cords
4. Treatment with another investigational drug or device within 30 days prior to signing Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being tested for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 6 months
  compare Sensitivity and Specificity to standard swab test

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Steady, MD, Principal Investigator — Soniphi LLC
Locations (1):
- Soniphi, Sebastopol, California, United States